CLINICAL TRIAL: NCT00432328
Title: A Double Blind, Placebo Controlled, Randomised Trial to Investigate the Efficacy of Juvista (Avotermin) in the Improvement of Scar Appearance in Patients Undergoing Bilateral Reduction Mammaplasty.
Brief Title: Juvista (Avotermin) in Breast Reduction Surgery Scars
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility analysis undertaken, determined that study was underpowered.
Sponsor: Renovo (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: RN1001-0041
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Mammaplasty; Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

INTERVENTIONS:
Drug: Avotermin

SUMMARY:
Severe scarring is a common problem following breast reduction surgery, studies have shown that over 64% of patients develop a hypertrophic scar at three months after the operation. Scar severity can be influenced by a large number of factors including age, sex, skin thickness and tension, ethnicity and the position of the scar on the body. Therefore the most sensitive and reliable method to assess the efficacy of an anti-scarring treatment is to compare bilateral wounds on the same individual. Bilateral breast reduction surgery provides an ideal model for a within patient evaluation of anti-scarring activity in wounds which develop into bad scars.

This study is being undertaken to investigate the efficacy and safety of Juvista (given as an intradermal injection of 200ng per 1cm wound margin) in the reduction of scar appearance applied to approximated wound margins following bilateral reduction mammaplasty.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 65 years of age undergoing bilateral reduction mammaplasty with anchor shaped incisions, who have given written informed consent.
* Patients with a Body Mass Index of 15-32 kg/m2 inclusive.
* Patients of child bearing potential who are using method(s) of contraception acceptable to the Investigator and agree to do so from at least the screening visit until 1 month after administration of the trial investigational products.
* Patients with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol.

Exclusion Criteria:

* Patients with significant breast asymmetry that may result in asymmetrical operative incisions being made on the left and rights breasts.
* Patients with breast asymmetry that may result in different post-operative tensions on the wounds of the left and right breasts.
* Patients who have had surgery in the area to be incised within one year of trial surgery.
* Patients with a history of a bleeding disorder.
* Patients with a history of breast malignancy.
* Patients with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the wounds or involves the areas to be examined in this trial.
* Patients who on direct questioning and/or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing.
* Patients with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Patients who are taking, or have taken, any investigational drugs in the 3 months prior to the screening visit.
* Patients who are taking regular, continuous, oral corticosteroid therapy.
* Patients undergoing investigations or changes in management for an existing medical condition.
* Patients who are or who become pregnant up to and including the day of surgery or who are lactating.
* Patients with diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety or efficacy of the investigational product.
* Patients who, in the opinion of the Investigator, are not likely to complete the trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Investigator scar assessment
Patient scar assessment
Independent scar assessment

SECONDARY OUTCOMES:
Local tolerance
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gilbert, FDSRCS FRCS, Principal Investigator — Queen Victoria Hospital, East Grinstead
Locations (6):
- United Kingdom (6):
  - Fitzwilliam Clinic, Belfast
  - Selly Oak Hospital, Birmingham
  - Queen Victoria Hospital, East Grinstead
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Preston Hospital, Preston
  - Odstock Centre for Burns & Plastic Surgery, Salisbury District Hospital, Salisbury